CLINICAL TRIAL: NCT04839679
Title: A Randomized Clinical Trial to Study the Utility of Visually Inspired Patient Education Material on Willingness to Pursue Radiation Therapy in American Indian and Alaska Native Individuals (VIEW Study)
Brief Title: A Study to Evaluate Visually Inspired Patient Education Material on Willingness to Pursue Radiation Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Samir Patel, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-005385; NCI-2021-13435 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Patient Education in Radiation Oncology
Keywords: Radiation therapy; Patient education; Radiation oncology; Native Americans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Mayo Clinic booklet (Active Comparator): Subjects will receive the standard Mayo Clinic educational booklet in preparation for clinically indicated radiation therapy treatment
  Interventions: Behavioral: Mayo Clinic Educational Booklet
- Culturally Oriented Education (Experimental): Subjects will receive a culturally appropriate educational brochure summarizing pertinent treatment information in a visual manner in addition to the standard Mayo Clinic booklet
  Interventions: Behavioral: Culturally Oriented Educational Brochure; Behavioral: Mayo Clinic Educational Booklet

INTERVENTIONS:
Behavioral: Culturally Oriented Educational Brochure — Culturally appropriate educational brochure summarizing pertinent treatment information in a visual manner
  Arms: Culturally Oriented Education
Behavioral: Mayo Clinic Educational Booklet — "An Introduction to Radiation Simulation and Treatment"- Barbara Woodward Lips, Patient Education Center

SUMMARY:
This research study is being done in order to better understand and identify American Indian/Alaskan Native (AI/AN) cancer patients' attitudes and beliefs towards radiation therapy treatment plans and their willingness to pursue them.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years of age with cancer diagnosis.
* Radiation therapy is recommended for their cancer treatment as a next step in their cancer care.
* Cognitive capacity to complete a paper-and-pencil survey.
* Ability to communicate and understand English with proficiency to provide informed consent and complete a paper-and-pencil survey.

Exclusion Criteria:

* Patient < 18 years of age.
* Patient does not have a cancer diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in patient anxiety | Baseline, day 14
  Measured using self-reported Hospital Anxiety and Depression Scale (HADS) Survey to ascertain any anxiety and/or depression that they may be experiencing with respect to their diagnosis and treatment. Questionnaire total score reported on a scale of 0-7 = normal, 8-10 borderline abnormal (borderline case), 11-21 abnormal (case)
Radiotherapy completion rates in the AI/AN community | 90 days
  Number of participates to complete radiation therapy as prescribed
Change in patient perception of information received | Baseline, day 14
  Measured by the EORTC QLQ - INFO25 survey, which is a validated instrument that will gauge their satisfaction with the information they received regarding their diagnosis and treatment plan. Questionnaire of 24 questions regarding information received during treatment using a scale of 1 (not at all) to 4 (very much).

CONTACTS AND LOCATIONS:
Overall Officials: Samir H. Patel, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials